CLINICAL TRIAL: NCT01616381
Title: Sildenafil in Heart Failure (SilHF); An Investigator Initiated Multinational Randomized Controlled Clinical Trial.
Brief Title: Sildenafil Versus Placebo in Chronic Heart Failure
Acronym: SilHF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SUS2011DIKE01; 2011-002829-21 (EudraCT Number)
Record Dates: First submitted 2012-06-01; First posted 2012-06-11 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Heart Failure; Pulmonary Hypertension
MeSH Terms: conditions — Heart Failure; Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sildenafil (Active Comparator): Sildenafil tablets 40 mg x 3 daily
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator): Placebo tablet x 3 daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — PDE-5 Inhibitor
  Other Names: Revatio
  Arms: Sildenafil
Drug: Placebo — Placebo for sildenafil 40mg x 3 daily
  Arms: Placebo

SUMMARY:
This protocol describes a 2-arm randomised controlled pilot study assessing the tolerance, safety and efficacy of sildenafil compared to control. The hypothesis is that sildenafil will be well tolerated and efficacious in patients with chronic heart failure (NYHA class II and III) with evidence of systolic dysfunction (EF ≤40 %) and secondary pulmonary hypertension (SPAP >40mmHg).

Patients that satisfy the inclusion criteria will be randomized to sildenafil (40mg x 3) or placebo therapy for 6 months in a 2:1 blinded fashion. The placebo group will be compared to the active therapy group and analysed for differences in the main study end-points Patient Global Assessment and 6-Minute Walk Test.

The study will also assess safety, tolerability, symptoms and quality of life.

DETAILED DESCRIPTION:
It is estimated that 2-3 % of the adult population suffers from heart failure (HF) and the prevalence is increasing. The European Society of Cardiology (ESC) represents countries with a population > 1,1 billion, and it is estimated that approximately 30 million patients have HF in these 53 countries. Heart failure is particularly prevalent in the elderly population and represents a major burden for both patients and the health services. HF is present in over 10% of patients admitted to hospital and accounts for ~ 2% of national health expenses. Approximately 50% of these costs are related to hospitalisation.

Despite optimal non-pharmacological, pharmacological and device therapy, the morbidity among HF patients is high with symptoms such as dyspnoea and fatigue that reduce quality of life. Following diagnosis approximately 50% are dead after 4 years. Forty percent of patients admitted to hospital with HF are either dead or rehospitalised within one year.

During the last decade, PDE5-inhibitors have been evaluated as a potential treatment for heart failure (see scientific rationale and reference). However, these investigations have been small and there is still limited data. Trials assessing the acute effects of PDE5-inhibition in patients with symptomatic HF due to systolic dysfunction have been performed primarily with sildenafil. Due to the short half-life of sildenafil the drug is administered 3 times daily when studying its chronic effects.

Previous studies have evaluated the 50 mg dose acutely and 50 mg 3 times daily during short-term chronic studies. Importantly, there is considerable off-label use of sildenafil in symptomatic heart failure patients in most European countries.

Revatio is currently licenced for pulmonary hypertension group 1. The dosing scheme is 20mg x 3. However, we suggest targeting a higher dose to achieve optimal clinical benefit in patients with heart failure and moderate congestion. As mentioned above most of the clinical literature in patients with symptomatic heart failure has been done using the 50mg x 3 regimen. However, it is believed that in the proposed study using 40mg x 3 should be equally efficacious. There is already considerable experience using this dosage scheme in heart failure patients locally.

The hemodynamic profile of PDE-5 inhibitors is favourable with reduction in filling pressures, both systemic and pulmonary, vascular resistance accompanied by improvement in symptoms and submaximal and peak exercise performance. This pilot study will evaluate the use of the PDE5-inhibitor sildenafil in patients with heart failure, systolic dysfunction and documented secondary pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women
2. 18 - 80 years of age.
3. Outpatients with chronic HF. NYHA class II-III on optimal treatment in sinus rhythm or atrial fibrillation
4. LVEF < 40% measured during the past 12 months
5. SPAP > 40mmHg using echocardiography
6. 6MWTD < 400 meters
7. NT-pro BNP > 400 pg/ml or BNP >100 pg/ml, measured during the past 12 months
8. Receiving optimal therapy, including diuretic, ACE-inhibitor, ARB, beta-blocker and aldosterone antagonist. Doses of all medication should be unchanged during the last 30 days before inclusion.
9. ICDs and CRTs (CRT-P, CRT-D) are permitted. Implantation should have been performed at > 3 months before inclusion to the trial.

Exclusion Criteria:

1. Acute Coronary Syndrome, including myocardial infarction, or coronary angiography, with or without intervention, within the last 3 months
2. Stroke within the last 3 months
3. Planned coronary angiography or planned device-implantation
4. Moderate to severe obstructive valve disease
5. Documented episodes of sustained ventricular tachycardia
6. Oral nitrate therapy or frequent use of sublingual nitrate
7. Concomitant disease which interfere with assessment of dyspnoea , severe COPD, asthma, restrictive lung disease, severe obesity
8. Anemia (hemoglobin < 10g/dL)
9. Uncontrolled hypertension ( SBP >160 mmHg and / or DBP > 90 mmHg)
10. Symptomatic or orthostatic hypotension or systolic blood pressure < 90 mmHg
11. Clinically important renal dysfunction (GFR < 40m ml/min)
12. Women with child-bearing potential
13. Use of

    i) alpha-1 antagonist: doxazosin

    ii) CYP3A4 inhibitors: erytromycin, ritonavir, sakinovir, itraconazole, ketoconazole

    iii) CYP3A4-inducers: rifampicin

    iv) Any calcium channel blockers
14. Retinitis pigmentosa, previous diagnosis of NAION (non-arteritic ischemic optic-neuropathy), unexplained visual disturbance.
15. Sickle cell anemia, multiple myeloma, leukemia or penile anatomic deformities (angulation, cavernosal fibrosis, Peyronie's disease) that increases the risk of priapism.
16. Hepatic failure.
17. Drug and alcohol abuse which precludes compliance with the protocol.
18. Inability to understand or sign the written informed consent form of the study,

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Patient Global Assessment | Baseline, 8 weeks, 24 weeks
  Analysis of change from baseline.
Six minute walk test | Baseline, 8 weeks, 24 weeks
  Analysis of change from baseline.

SECONDARY OUTCOMES:
Quality of Life (QoL) evaluation by EuroQol5D | Baseline, 8 weeks and 24 weeks
  Analysis of change from baseline.
Kansas City Questionaire | Baseline, 8 weeks and 24 weeks
  Analysis of change from baseline.
New York Heart Association (NYHA) function class | Baseline, 8 weeks, 16 weeks and 24 weeks
  Analysis of change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Dickstein, MD, PhD, Principal Investigator — Helse Stavanger HF
Locations (6):
- Israel (2):
  - Lady Davis Carmel Medical CEnter, Haifa
  - Rabin Medical Center, Petah Tikva
- San Donato Hospital, Milan, Italy
- Stavanger University Hospital, Stavanger, Rogaland, Norway
- United Kingdom (2):
  - Castle Hill Hospital, Hull
  - Northern General Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooper TJ, Guazzi M, Al-Mohammad A, Amir O, Bengal T, Cleland JG, Dickstein K. Sildenafil in Heart failure (SilHF). An investigator-initiated multinational randomized controlled clinical trial: rationale and design. Eur J Heart Fail. 2013 Jan;15(1):119-22. doi: 10.1093/eurjhf/hfs152. Epub 2012 Oct 24. PMID 23097067